CLINICAL TRIAL: NCT02678403
Title: Efficacy of Transcutaneous Electrical Nerve Stimulation in the Improvement of Walking Distance in Patients With Peripheral Artery Disease With Intermittent Claudication
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation in Peripheral Artery Disease TENS-PAD Study / TENS-AOMI
Acronym: TENS-PAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: principal investigator left Toulouse hospital
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/14/7386; 2015-A01534-45 (Other: ID-RCB)
Record Dates: First submitted 2016-01-08; First posted 2016-02-09 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; transcutaneous electrical nerve stimulation; walking ability; endothelial function
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - TENS group (Experimental): The treatment will consist of Transcutaneous electrical nerve stimulation (TENS): stimulation of the leg (frequency of 10 Hz, Biphasic, with a pulse width of 200 µs, maximal intensity below motor threshold), 45 minutes per day, in the morning before the exercise rehabilitation programme, for 3 weeks, 5 days per week.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- 2 - SHAM group (Sham Comparator): SHAM Transcutaneous electrical nerve stimulation (TENS) : the stimulation placebo will be delivered according to the same modalities as for the TENS group but with a voltage level that vanishes automatically after 10 seconds of stimulation.
  Interventions: Device: SHAM Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) is the use of electric current produced by a device to stimulate the nerves that only induces sensory stimulation (without muscle contraction) and is classically used in the treatment of pain.
  Arms: 1 - TENS group
Device: SHAM Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) is the use of electric current produced by a device to stimulate the nerves that only induces sensory stimulation (without muscle contraction) and is classically used in the treatment of pain.
  Arms: 2 - SHAM group

SUMMARY:
Purpose: The investigators team recently carried out a proof of concept study testing the efficacy of one single 45-minute session of 10 Hz TENS prior to walking, versus placebo. In this randomized study, the investigators found that TENS significantly delayed pain onset and increased the pain-free walking distance in patients with class II PAD. From these encouraging results, the investigators now seek to assess the efficacy of an intervention that includes the daily use of TENS for 3 weeks (5 days a week) on walking distance in PAD (Leriche-Fontaine stage II). Methods/Design: prospective multicentre study / randomized controlled trial / double blinding.

DETAILED DESCRIPTION:
Interventions (2 groups): Experimental group (TENS group): the treatment will consist of stimulation of the leg (frequency of 10 Hz, Biphasic, with a pulse width of 200 µs, maximal intensity below motor threshold), 45 minutes per day, in the morning before the exercise rehabilitation programme, for 3 weeks, 5 days per week. Control group (group SHAM): the stimulation placebo will be delivered according to the same modalities as for the TENS group but with a voltage level that vanishes automatically after 10 seconds of stimulation.

15 days of interventions (TENS or SHAM) between J0 and J23, End of study for patient at J24-J25, two days for the last analyses who are the same of inclusion's visit J0.

Primary outcome: walking distance (metres) measured on a treadmill with a standardized protocol. Secondary outcomes: transcutaneous oxygen pressure (TcPO2) measured during a Strandness exercise test, peak oxygen uptake (VO2 peak) (ml.min.kg-1), endothelial function (EndoPAT®), ankle-brachial pressure index, body mass index, lipid profile (LDL-C, HDL-C, Triglycerides), fasting glycaemia, HbA1c, WELCH questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Leriche stage II PAD, admitted to cardiovascular Rehabilitation Unit
* Men or women
* Able to take part in an out-patient rehabilitation programme
* Clinically stable
* Sedentary
* Provided informed consent to participate in the study

Exclusion Criteria:

* Ward of court
* Walking disorders related to orthopaedic or neuromuscular disease
* Participation in a structured physical reconditioning programme in the month before the study
* Renal insufficiency requiring dialysis
* Known and documented myopathy
* Progressive cancer
* Associated progressive disease causing a deterioration in general health
* Participation in another research protocol
* Skin disorder making it impossible to use TENS
* Absolute contra-indication to physical activity
* Presence of pacemaker / defibrillator
* Pregnant women in the 1st trimester / 12 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
walking distance without pain (in meters) | Change between J0 and J25 (15 days)
  the evolution of the claudication distance between the start and the end of the study (1 session of TENS each day , 15 days in total) in the two intervention group (TENS vs SHAM). Measure of change between inclusion and end of study.

SECONDARY OUTCOMES:
maximal oxygen consumption (VO2peak in ml.min) | Change between J0 and J25 (15 days)
  maximal oxygen consumption (VO2peak in ml.min) Measure of change between inclusion and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Marc LABRUNEE, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - University Hospital of Dijon, Dijon
  - University Hospital of Nîmes, Nîmes
  - Clinique de Saint-Orens, Saint-Orens-de-Gameville
  - Toulouse University Hospital (CHU de Toulouse), Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besnier F, Senard JM, Gremeaux V, Riedel M, Garrigues D, Guiraud T, Labrunee M. The efficacy of transcutaneous electrical nerve stimulation on the improvement of walking distance in patients with peripheral arterial disease with intermittent claudication: study protocol for a randomised controlled trial: the TENS-PAD study. Trials. 2017 Aug 10;18(1):373. doi: 10.1186/s13063-017-1997-1. PMID 28797281